CLINICAL TRIAL: NCT02033291
Title: Blood-Brain Barrier Permeability Quantification in Cerebral Small Vessel Disease -- Reproducibility of Dynamic Contrast-enhanced MRI
Brief Title: Blood-brain Barrier Quantification in Cerebral Small Vessel Disease
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 13-2-036
Record Dates: First submitted 2014-01-08; First posted 2014-01-10 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Blood-Brain Barrier Permeability; Cerebral Small Vessel Disease; Cerebral Hemorrhage; Cortical Stroke
Keywords: Cerebral Small Vessel Disease; Blood-Brain Barrier permeability; Dynamic contrast enhanced Magnetic Resonance Imaging; Pharmacokinetic modeling; Reproducibility
MeSH Terms: conditions — Cerebral Small Vessel Diseases; Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cortical stroke or primary intracerebral hemorrhage patients:: patients who have a clear clinical presentation of either cortical stroke or primary intracerebral hemorrhage confirmed on brain CT. The patients are eligible when the DCE-MRI scans can be performed within 0-6 weeks of the vascular event and on two subsequent days as the vascular permeability may change significantly on the timescale of weeks.
  Interventions: Procedure: Dynamic contrast enhanced Brain MRI
- cSVD patients: patients who present with a transient ischemic attack (TIA) and cSVD related abnormalities on brain MRI. TIA patients are defined as patients with stroke like symptoms that last no longer than 24 hours. MRI abnormalities include extended white matter lesions, (asymptomatic) lacunar infarcts, microbleeds and enlarged Virchow-Robin spaces. The patients are eligible when the first DCE-MRI scan can be performed 8-12 weeks after the TIA to avoid the acute phase, and the second MRI-scan within four weeks after the first.
  Interventions: Procedure: Dynamic contrast enhanced Brain MRI

INTERVENTIONS:
Procedure: Dynamic contrast enhanced Brain MRI — DCE-MRI is used to quantify the BBB permeability

SUMMARY:
Cerebral small vessel disease (cSVD) encompasses all pathological processes that affect the small vessels of the brain. On brain-MRI cSVD is characterized by structural brain abnormalities such as white matter lesions (WMLs). Clinically, cSVD is related to acute syndromes as lacunar stroke but also to more chronic health problems such as cognitive decline. Recent literature suggests that a disrupted blood brain barrier (BBB), leading to elevated BBB permeability, may play a pivotal role in the aetiology of cSVD and lacunar stroke. The BBB is a complex system of neuronal, glial and vascular cells which main function is to shield the brain from toxic components and regulate the homeostasis. Elucidating the role of the BBB may have far reaching consequences for the treatment of cSVD patients and the reduction of recurrence rate of the disease. This could lead to a better quality of life among cSVD patients and reduce the economic burden on society. Currently the exact contribution and extent of a possibly defective BBB in cSVD remains largely unclear, due to the lack of a reliable method to accurately quantify the BBB permeability in cSVD patients. As a result, the current treatment consists of treating the cardiovascular risk factors, often with poor results.

Quantification of the BBB permeability provides an objective measure of the integrity of the BBB and as such aids the study of the role of the BBB. The aim of this study is to realize a clinically applicable MRI-method to quantify the BBB permeability. Moreover, the method can be used to study the involvement of BBB disruption in other neuropathologies including Alzheimer's disease, vascular dementia, hypertension and diabetes.

Primary Study Objective:

To realize a clinically applicable quantification of BBB permeability using DCE-MRI by determining the reproducibility of the DCE-MRI method

Secondary Study Objective:

To achieve the shortest scan duration without compromising the reliability of the BBB permeability quantification.

Hypotheses:

1. Using an optimized DCE-MRI method to quantify the BBB permeability, the BBB permeability can be reliably determined in cSVD patients.
2. The scan duration can be shortened without compromising the reliability of the BBB permeability quantification.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

* Age >18 years old
* The condition of the patient must be well enough to allow participation in the study, which is decided in consultation with the treating physician.

cSVD patients: - patients who present with a transient ischemic attack (TIA) and cSVD related abnormalities on brain MRI. TIA patients are defined as patients with stroke like symptoms that last no longer than 24 hours. MRI abnormalities include extended white matter lesions, (asymptomatic) lacunar infarcts, microbleeds and enlarged Virchow-Robin spaces. The patients are eligible when the first DCE-MRI scan can be performed 8-12 weeks after the TIA to avoid the acute phase, and the second MRI-scan within four weeks after the first.

Cortical stroke or primary intracerebral hemorrhage patients:

- patients who have a clear clinical presentation of either cortical stroke or primary intracerebral hemorrhage confirmed on brain CT. The patients are eligible when the DCE-MRI scans can be performed within 0-6 weeks of the vascular event and on two subsequent days as the vascular permeability may change significantly on the timescale of weeks.

Exclusion Criteria:

All subjects:

* History of cerebrovascular disease (e.g. ischemic/hemorrhagic stroke)
* History of other diseases of the central nervous system (e.g. epilepsy, brain tumor, multiple sclerosis)
* Contra-indications for MRI examination: e.g. pacemaker; neurostimulator; medication pump; cochlear or hearing implant; tattoos or other items that cannot be removed and include metal parts (for instance from operations in the past); metal splinter in the eye; pregnancy and claustrophobia; brain vessel clamps; denture, which contains magnets.
* Contra-indication for MRI contrast agent: e.g. strong suspicion for impaired kidney function (GFR<30ml/min), previous allergic reaction to contrast agent, dialysis patients
* Psychiatric co-morbidity and inability to perform the (DCE-)MRI scans.

cSVD patients

* Patients with a potential cardioembolic source (e.g. atrial fibrillation)
* Stenosis of ≥50% of one or both internal carotid arteries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General:
  * Age >18 years old
  * The condition of the patient must be well enough to allow participation in the study, which is decided in consultation with the treating physician.
  cSVD patients: - patients who present with a transient ischemic attack (TIA) and cSVD related abnormalities on brain MRI. MRI abnormalities include extended white matter lesions, (asymptomatic) lacunar infarcts, microbleeds and enlarged Virchow-Robin spaces. The patients are eligible when the first DCE-MRI scan can be performed 8-12 weeks after the TIA to avoid the acute phase, and the second MRI-scan within four weeks after the first.
  Cortical stroke or primary intracerebral hemorrhage patients:
  - patients who have a clear clinical presentation of either cortical stroke or primary intracerebral hemorrhage confirmed on brain CT. The patients are eligible when the DCE-MRI scans can be performed within 0-6 weeks of the vascular event and on two subsequent days.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2014-02; Primary Completion 2015-12 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
pharmacokinetic parameter values Ki and vb | day 1 & day 2. Day 2 is min. 24 hours max. 4 weeks after day 1.
  Outcome measures of both days are used to determine the reproducibility of the DCE-MRI method.

SECONDARY OUTCOMES:
pharmacokinetic parameter values: Ki and vb for the retrospectively shortened dynamic scans | Day 1
  The pharmacokinetic parameters are evaluated as a function of scan duration to obtain the shortest scan duration without compromising the reliability of the BBB permeability quantification.

CONTACTS AND LOCATIONS:
Overall Officials: Cecile RLPN Jeukens, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands